CLINICAL TRIAL: NCT05038241
Title: HORMONAL ROLE IN VERNAL KERATOCONJUNCTIVITIS
Brief Title: HORMONES IN VERNAL KERATOCONJUNCTIVITIS
Acronym: HOR-VKC-2020
Status: Completed | Type: Observational
Sponsor: Fondazione IRCCS Ca' Granda, Ospedale Maggiore Policlinico (Other)
Responsible Party: Sponsor
Other Study IDs: 1965
Record Dates: First submitted 2021-08-29; First posted 2021-09-09 (Actual); Last update posted 2022-04-22 (Actual); Status verified 2021-08

CONDITIONS: Conjunctivitis, Vernal
MeSH Terms: conditions — Conjunctivitis, Allergic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Active VKC: All females and males of pubertal age with active VKC undergo a blood sample for the determination of serum hormone levels, an allergological evaluation and an endocrinological evaluation. All is done at the time of enrollment.
- Previous active VKC: All females and males of pubertal age who suffered of VKC undergo a blood sample for the determination of serum hormone levels, an allergological evaluation and an endocrinological evaluation. All is done at the time of enrollment.

SUMMARY:
VKC is more common in males and tends to resolve with pubertal development. Clinical observation was not followed by an investigation that clarified whether there is a correlation between the hormonal pattern and the evolution of the disease, in particular it is not defined whether there is a correlation between the hormonal pattern and the resolution of the disease.

This study aims to evaluate the hormonal pattern in patients with VKC and, in particular, the possible role of these hormones in the resolution of this condition in puberty.

DETAILED DESCRIPTION:
The study presents a retrospective and prospective transversal observational design, non-pharmacological, monocentric, non-profit.

It is based on the collection of clinical, laboratory and therapy data on databases of patients affected by Vernal keratoconjunctivitis.

Participation in the study will be proposed to parents of patients with VKC over 10 years of age at puberty (B2 according to Tanner for females and G2 according to Tanner for males), based on endocrinological evaluation. Patients, differentiated by gender, will be divided into two groups: patients with active VKC and patients with resolved VKC. Both study groups will be offered a blood sample to determine the serum levels of LH, FSH, estradiol, DHEAS, androstenedione, total testosterone, SHBG, DHT, 17OH-progesterone, TSH-R, albumin, ACTH and cortisol. In postpuberal females, the sample must be taken in the first 5 days of the menstrual cycle.

This study provides for the enrollment of patients diagnosed with VKC followed at the Allergy Outpatient Clinic of the UOSD Pediatrics High Intensity of Care - IRCCS Ca 'Granda Foundation Ospedale Maggiore Policlinico di Milano. The source documentation of the data will be the medical record and the reports of the examinations, provided for by the study, performed at the Institute. On the same day, a blood sample and a pubertal stage assessment will be performed. An allergy / ophthalmological examination for VKC will be carried out only if it had not been performed in the 12 months prior to the execution of the blood sample. There is no follow-up.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of VKC assessed by an allergologist or ophthalmologist over 10 years of age

Exclusion Criteria:

* Presence of pre-existing pathologies of the endocrine system.

Ages: 10 Years to 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: The study involves the enrollment of 2 groups of subjects: pubertal patients with active VKC and pubertal / postpuberal patients who have suffered from VKC in the past years, but no longer in 2021. To all the subjects under examination, both males both females, a blood sample is performed for the determination of hormonal levels, an allergological / ophthalmological evaluation to determine the phase of activity of the VKC and an endocrinological evaluation to determine the degree of pubertal development.
Sampling Method: Non-Probability Sample
Enrollment: 88 (Actual)
Dates: Start 2021-04-01 (Actual); Primary Completion 2021-10-31 (Actual); Study Completion 2021-12-31 (Actual)

PRIMARY OUTCOMES:
To assess the difference in serum total testosterone levels between the population of subjects with active VKC and the population of subjects with resolved VKC. | All subjects enrolled between April 2021 and October 2021 undergo a venous blood sample for the determination of plasma testosterone. This withdrawal is made in the morning, between 8.30 and 9.30 am, in a single determination at the time of enrollment.
  A venous blood sample is taken from all enrolled subjects for the determination of plasma testosterone. This collection is made in the morning, between 8.30 and 9.30 am.

SECONDARY OUTCOMES:
To evaluate the difference in serum levels of the other hormones investigated between the population of subjects with active VKC and the population of subjects with resolved VKC. | All subjects enrolled between April 2021 and October 2021 undergo a venous blood sample for the determination of plasma hormones. This withdrawal is made in the morning, between 8.30 and 9.30 am, in a single determination at the time of enrollment.
  A venous blood sample is taken from all enrolled subjects for the determination of hormones. This collection is made in the morning, between 8.30 and 9.30 am.
To assess the correlation between serum hormone levels and VKC activity. | All subjects enrolled between April 2021 and October 2021 undergo a venous blood sample for plasma hormones. This withdrawal is made in the morning, between 8.30 and 9.30 am, in a single determination at the time of enrollment.
  A venous blood sample is taken from all enrolled subjects for the determination of plasma hormones. This collection is made in the morning, between 8.30 and 9.30 am. VKC activity is determined by an allergologic evaluation at the time of enrollment.
To evaluate the possible presence of a serum hormone marker that may be related to the resolution of ocular symptoms. | All subjects enrolled between April 2021 and October 2021 undergo a venous blood sample for plasma hormones. This withdrawal is made in the morning, between 8.30 and 9.30 am, in a single determination at the time of enrollment.
  A venous blood sample is taken from all enrolled subjects for the determination of plasma hormones. This collection is made in the morning, between 8.30 and 9.30 am. VKC activity is determined by an allergologic evaluation at the time of enrollment.

CONTACTS AND LOCATIONS:
Locations (1):
- dr. Daniele Giovanni Ghiglioni, Milan, Italy